CLINICAL TRIAL: NCT01555073
Title: A Prospective Randomized Blinded Placebo Controlled Comparison of Multimodal Pre-emptive Analgesia on Long Term Outcome Following Uterine Artery Embolization
Brief Title: Preemptive Analgesia Following Uterine Artery Embolization
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subjects did not meet inclusion criteria
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor in Anesthesiology and Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00004604
Record Dates: First submitted 2011-10-14; First posted 2012-03-15 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Uterine Fibroids; Uterine Artery Embolization
MeSH Terms: conditions — Leiomyoma | interventions — Pregabalin; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin/celecoxib group (Active Comparator): pregabalin/celecoxib twice a day for 13 days.
  Interventions: Drug: pregabalin/celecoxib
- Pregabalin/placebo group (Active Comparator): pregabalin/placebo twice a day for 13 days.
  Interventions: Drug: pregabalin/placebo
- Celecoxib/placebo group (Active Comparator): celecoxib/placebo twice a day for 13 days.
  Interventions: Drug: celecoxib/placebo
- Placebo group (Placebo Comparator): Placebo group, two placebo tablets day of surgery and twice a day for 13 days
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: pregabalin/celecoxib — pregabalin/celecoxib; 75mg/400mg day of surgery and (75mg/200mg) twice a day for 13 days.
  Other Names: Celebrex; Lyrica
  Arms: Pregabalin/celecoxib group
Drug: pregabalin/placebo — pregabalin/placebo; 75mg/placebo day of surgery and (75mg/placebo) twice a day for 13 days.
  Other Names: Lyrica
  Arms: Pregabalin/placebo group
Drug: celecoxib/placebo — celecoxib/placebo; 400mg/placebo day of surgery and 200mg/placebo twice a day for 13 days.
  Other Names: Celebrex
  Arms: Celecoxib/placebo group
Drug: Placebo group — Placebo group, two placebo tablets day of surgery and twice a day for 13 days
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
Uterine leiomyomata, also known as fibroids, are an extremely common benign lesion being present in 30-50% of all women. Traditional surgical treatment of symptomatic fibroids has been hysterectomy in post child bearing woman. However, over the last decade, the use of a minimal invasive technique called uterine artery embolization has become increasingly popular due to high patient satisfaction, cost effectiveness, and shorter recovery period. The purpose of this randomized blinded placebo controlled study is to compare pre-emptive analgesia vs non-preemptive analgesia for immediate postoperative pain control, long term pain control, and improved quality of life in woman following uterine artery embolization surgery. The study consists of four drug groups including a placebo group. The addition of pregabalin and celecoxib together with epidural analgesia may improve pain management as well as leading to a better post-procedure outcome in women following uterine artery embolization.

Many investigators believe that the ischemia in the normal myometrium is the primary source of pain immediately following surgery making postoperative pain management challenging. Epidural fentanyl may offer an advantage when encountering visceral pain. In addition to being an effective analgesic for chronic pain syndromes, the use of pregabalin provides effective postoperative analgesia when it is administered pre-emptively before an operation. Preemptive analgesia involves the introduction of an analgesic regimen before the onset of noxious stimuli, with the goal of preventing sensitization of the nervous system to subsequent stimuli that could amplify pain. In human trials, pregabalin has been demonstrated to reduce pain, improve sleep, and mood disturbances in patients with post herpetic neuralgia. The use of celecoxib in combination with pregabalin has shown to provide more effective analgesia by providing antihyperalgesia. Therefore, the addition of pregabalin and celecoxib together with epidural analgesia may improve pain management as well as having an effect on long term sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients (>18 years of age) who are undergoing elective uterine artery embolization will be included in the study.

Exclusion Criteria:

* Exclusion criteria for the study are patient refusal to be included in the study, the presence of language barrier that inhibits proper communication with the patient
* Contraindications to regional anesthesia
* History of allergy to amide local anesthetics or narcotics
* Known hypersensitivity to pregabalin, creatinine clearance ≤ 60 mL/min
* The presence of a progressive neurological deficit
* The presence of chronic opioid analgesia
* The presence of a coagulopathy or infection, pregnancy
* Patients with cardiovascular disease
* Patients who take daily antiplatelet medications, patients with peptic ulcer disease
* History of psychiatric disorder or inability to follow study protocol.
* Dropout criteria include failed epidural analgesia, inability to tolerate side effects (nausea) from pregabalin, and the inability to contact during follow up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin/Celecoxib Group | Pregabalin/Placebo Group | Celecoxib/Placebo Group | Placebo Group
Started | 7 | 3 | 7 | 6
Completed | 6 | 1 | 7 | 1
Not Completed | 1 | 2 | 0 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Baseline Analysis population description
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin/Celecoxib Group | Pregabalin/Placebo Group | Celecoxib/Placebo Group | Placebo Group | Total
Number analyzed (Participants) | 7 | 3 | 7 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 7 | 6 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 7 | 6 | 23
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain Control
Description: To evaluate the post operative pain control of the four groups in immediate postoperative period and months following uterine artery embolisation procedure.
Time Frame: Expected average of 12 weeks
Population: Early termination due to lost of follow-up for primary outcome at 3 months
Arm/Group | Pregabalin/Celecoxib Group | Pregabalin/Placebo Group | Celecoxib/Placebo Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Quality of Life
Description: To register the quality of life of patients receiving the four study arms following uterine artery embolisation during immediate and long term time periods.
Time Frame: Expected average of 12 weeks
Population: Early termination due to lost of follow-up for primary outcome at 3 months
Arm/Group | Pregabalin/Celecoxib Group | Pregabalin/Placebo Group | Celecoxib/Placebo Group | Placebo Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pregabalin/Celecoxib Group | Pregabalin/Placebo Group | Celecoxib/Placebo Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/3 | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Early termination due to lost of follow-up for primary outcome at 3 months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes